CLINICAL TRIAL: NCT03225508
Title: A Novel Method to Measure Diaphragmatic Motion and Excursion
Brief Title: Diaphragmatic Motion Using Linear Ultrasound
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 16-6385
Record Dates: First submitted 2017-07-19; First posted 2017-07-21 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Diaphragm; Movement; Examination of Diaphragm Movement Using Ultrasound
MeSH Terms: interventions — Respiratory Function Tests

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Phase 1: The first phase will be to evaluate a new lung ultrasound technique to measure diaphragmatic excursion using a linear probe in the mid-axillary line. This will involve scanning 75 healthy patients undergoing elective surgery to determine normal reference values in men and women.
  The following interventions will be carried out:
  (i) Measurement of diaphragmatic movement with a linear ultrasound probe on both sides of the chest (ii) Measurement of diaphragmatic movement with a curved ultrasound probe on both sides of the chest
  Interventions: Diagnostic Test: Linear Ultrasound to Measure Diaphragmatic Movement; Diagnostic Test: Curvilinear Ultrasound to Measure Diaphragmatic Movement
- Phase 2: This will involve patients undergoing an interscalene / supraclavicular brachial plexus block for their routine care, it will examine the reduction in diaphragmatic motion due to phrenic nerve palsy.
  Interventions:
  (i) Measurement of diaphragmatic movement with a linear ultrasound probe bilaterally.
  (ii) Measurement of diaphragmatic movement with a curved ultrasound probe bilaterally.
  (iii) Pulmonary function tests prior to the brachial plexus block (iv) Planned supraclavicular / interscalene block by the clinical team. (v) Repeat measurement of diaphragmatic movement with linear ultrasound, only on the side of the brachial plexus block.
  (vi) Repeat measurement of diaphragmatic movement with curved ultrasound, only on the side of the brachial plexus block.
  Interventions: Diagnostic Test: Linear Ultrasound to Measure Diaphragmatic Movement; Diagnostic Test: Curvilinear Ultrasound to Measure Diaphragmatic Movement; Diagnostic Test: Pulmonary function tests

INTERVENTIONS:
Diagnostic Test: Linear Ultrasound to Measure Diaphragmatic Movement — A linear 10-12 MHz ultrasound probe will be used to determine diaphragmatic excursion, by examining the zone of apposition. Diaphragmatic excursion will be measured from end inspiration to end expiration. The measurement will be repeated twice, and an average of the two will be taken. The distance between the two external skin markings, one at the end of full expiration and one at the end of full inspiration will indicate the excursion of the diaphragm.
Diagnostic Test: Curvilinear Ultrasound to Measure Diaphragmatic Movement — A curvilinear 2-5 MHz ultrasound probe will be used to determine diaphragmatic excursion, by examining the dome of the diaphragm. M-mode will be used to image the motion of the diaphragm from end inspiration to end expiration. The measurement will be repeated twice, and an average of the two will be taken.
Diagnostic Test: Pulmonary function tests — Bedside pulmonary function tests to measure forced vital capacity (FVC). The FVC measures the maximal volume of gas that can be expired as forcefully and rapidly as possible after a maximal inspiration to total lung capacity. This measurement will help determine if the patient has any obstructive or restrictive diseases of the airways. Three measurements will be taken.
  Groups: Phase 2

SUMMARY:
This study evaluates the movement of the diaphragm (which is the main muscle used for breathing). It will compare two ultrasound modalities: linear ultrasound versus curvilinear ultrasound, at measuring diaphragm motion. The proposed measurement method with linear ultrasound is novel, and will be compared against the established method with curvilinear ultrasound. The investigators hypothesize that the novel method will have several potential advantages, including: it may be easier to learn, quicker to perform, and have a lower failure rate.

DETAILED DESCRIPTION:
Background:

Multiple pathologies cause diaphragmatic dysfunction, including: respiratory, abdominal and neurological disease. Established clinical tests of diaphragmatic function, include: the transdiaphragmatic pressure, the maximal static inspiratory pressure, the sniff inspiratory pressure, pulmonary function tests, electromyography, a chest radiograph or fluoroscopy.

However ultrasound assessment of diaphragmatic function is a non-invasive, radiation-free technique that has gained traction in clinical practice in recent years. Several different methods have been described, that examine motion in two different areas of the diaphragm, either the zone of apposition, or the dome of the diaphragm, however no one method has emerged as the standard of care.

The current conventional technique (using B-mode or M-mode ultrasound via a phased array or curvilinear probe) in the subcostal region, has several limitations:

* It can be difficult to measure right hemi-diaphragm excursion with deep breathing, with a failure rate of up to 28% described for quantitative assessment.
* It is even more difficult to quantitatively assess left hemi-diaphragmatic excursion with deep breathing, as the spleen provides a smaller window compared to the liver window. Failure rates of 79% and 65% have been reported.
* When using M-mode, the ultrasound beam must image the diaphragmatic excursion line at a perpendicular angle, otherwise reproducibility and accuracy are adversely effected.

The investigators propose a novel method, using linear ultrasound to examine the zone of apposition, and determine diaphragmatic excursion at end inspiration and expiration. In theory this technique may have a number of advantages over the conventional method. It is likely easier to learn, quicker to perform, and has a lower failure rate for imaging the diaphragm on both sides during deep breathing. The investigators will compare this method to the conventional method, i.e. a curvilinear probe as described above.

Hypothesis:

Diaphragmatic motion can be assessed more rapidly, and more reliably via a linear high frequency ultrasound probe, than a curved low frequency probe.

Primary Objective:

- To evaluate the ease and success of using a novel technique of point-of-care ultrasound diaphragm assessment with a linear probe in the mid-axillary line to measure diaphragmatic motion. The ease of procedure will be determined by the time and the number of attempts required to perform the ultrasound assessment.

Secondary Objectives:

* To determine the normal range of diaphragmatic excursion values from full expiration to full inspiration in men and women;
* To quantify the reduction in diaphragmatic motion following phrenic nerve palsy - due to an interscalene, upper trunk or supraclavicular brachial plexus block;
* To compare the finding of diminished diaphragmatic excursion with the conventional method of measurement; i.e. compare the sensitivity and specificity of the tests.
* To analyze the success rate of measuring the left and right hemi-diaphragmatic movement as compared with the conventional method of measurement.

This prospective observational study, will involve patients undergoing elective surgery, and will consist of two phases:

Phase 1:

The first phase will be to evaluate a new lung ultrasound technique to measure diaphragmatic excursion using a linear probe in the mid-axillary line. This will involve scanning 75 healthy patients undergoing elective surgery to determine normal reference values for this technique in men and women.

Phase 2:

The second phase will involve 100 patients who are undergoing an inter-scalene, upper trunk of cervical plexus, or supraclavicular brachial plexus block as part of their perioperative analgesic management for shoulder or arm surgery. This cohort of patient is likely to develop phrenic nerve palsy as a side effect of the brachial plexus block. The resultant phrenic nerve palsy, will result in reduced diaphragmatic motion, and the aim will be to evaluate the ability of using a linear probe technique to measure this reduction as compared to the conventional method of measurement.

ELIGIBILITY:
Inclusion Criteria:

Phase 1 Any healthy adult patient undergoing elective surgery

Phase 2 Any adult patient, undergoing elective upper limb surgery that involves an interscalene or supraclavicular brachial plexus block.

Exclusion Criteria:

(i) Inability to obtain an informed consent (e.g. language barrier) (ii) BMI > 35 (iii) Known pre-existing diaphragmatic dysfunction (iv) Existing lung pathology

1. Smoker
2. Known abnormal pulmonary function tests
3. Severe pulmonary disease e.g., COPD, asthma, pulmonary fibrosis, or any other significant respiratory disease that would adversely affect diaphragm function or pulmonary function tests

Additional Criteria for Phase 2 Any contraindication to an interscalene or supraclavicular brachial plexus block

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Phase 1 Any healthy adult patient undergoing elective surgery
  Phase 2 Any adult patient, undergoing elective upper limb surgery that involves an interscalene or supraclavicular brachial plexus block.
Sampling Method: Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2017-06-09 (Actual); Primary Completion 2024-05-23 (Actual); Study Completion 2024-05-23 (Actual)

PRIMARY OUTCOMES:
Time taken to measure diaphragmatic excursion | 60 minutes
  To measure in minutes the time taken to quantify diaphragmatic excursion from end inspiration to end expiration, and to compare the linear probe versus the curvilinear probe.

SECONDARY OUTCOMES:
Normal range of values for diaphragmatic excursion using linear ultrasound | 30 mins
  To determine the normal range of values for diaphragmatic excursion from end expiration to end inspiration in men and women
Quantify and compare the reduction in diaphragmatic motion following a phrenic nerve block | 2 hours
  To quantify and compare the reduction in diaphragmatic motion (% change from baseline) following a phrenic nerve block using both linear and curved ultrasound probes
Success rate of measuring both the left and right hemi-diaphragmatic movement | 60 mins
  To analyze the success rate of measuring both the left and right hemi-diaphragmatic movement; success is defined as successful capture of a good view of the diaphragm and its movement on sonogram using the B mode and M mode scan

CONTACTS AND LOCATIONS:
Overall Officials: Anahi Perlas, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sferrazza Papa GF, Pellegrino GM, Di Marco F, Imeri G, Brochard L, Goligher E, Centanni S. A Review of the Ultrasound Assessment of Diaphragmatic Function in Clinical Practice. Respiration. 2016;91(5):403-11. doi: 10.1159/000446518. Epub 2016 May 25. PMID 27216909
- [Background] Boussuges A, Gole Y, Blanc P. Diaphragmatic motion studied by m-mode ultrasonography: methods, reproducibility, and normal values. Chest. 2009 Feb;135(2):391-400. doi: 10.1378/chest.08-1541. Epub 2008 Nov 18. PMID 19017880
- [Background] Kim SH, Na S, Choi JS, Na SH, Shin S, Koh SO. An evaluation of diaphragmatic movement by M-mode sonography as a predictor of pulmonary dysfunction after upper abdominal surgery. Anesth Analg. 2010 May 1;110(5):1349-54. doi: 10.1213/ANE.0b013e3181d5e4d8. PMID 20418298
- [Background] Kim WY, Suh HJ, Hong SB, Koh Y, Lim CM. Diaphragm dysfunction assessed by ultrasonography: influence on weaning from mechanical ventilation. Crit Care Med. 2011 Dec;39(12):2627-30. doi: 10.1097/CCM.0b013e3182266408. PMID 21705883
- [Background] Lerolle N, Guerot E, Dimassi S, Zegdi R, Faisy C, Fagon JY, Diehl JL. Ultrasonographic diagnostic criterion for severe diaphragmatic dysfunction after cardiac surgery. Chest. 2009 Feb;135(2):401-407. doi: 10.1378/chest.08-1531. Epub 2008 Aug 27. PMID 18753469
- [Background] Testa A, Soldati G, Giannuzzi R, Berardi S, Portale G, Gentiloni Silveri N. Ultrasound M-mode assessment of diaphragmatic kinetics by anterior transverse scanning in healthy subjects. Ultrasound Med Biol. 2011 Jan;37(1):44-52. doi: 10.1016/j.ultrasmedbio.2010.10.004. PMID 21144957
- [Background] Baldwin CE, Paratz JD, Bersten AD. Diaphragm and peripheral muscle thickness on ultrasound: intra-rater reliability and variability of a methodology using non-standard recumbent positions. Respirology. 2011 Oct;16(7):1136-43. doi: 10.1111/j.1440-1843.2011.02005.x. PMID 21645172
- [Background] DiNino E, Gartman EJ, Sethi JM, McCool FD. Diaphragm ultrasound as a predictor of successful extubation from mechanical ventilation. Thorax. 2014 May;69(5):423-7. doi: 10.1136/thoraxjnl-2013-204111. Epub 2013 Dec 23. PMID 24365607
- [Background] Ferrari G, De Filippi G, Elia F, Panero F, Volpicelli G, Apra F. Diaphragm ultrasound as a new index of discontinuation from mechanical ventilation. Crit Ultrasound J. 2014 Jun 7;6(1):8. doi: 10.1186/2036-7902-6-8. eCollection 2014. PMID 24949192
- [Background] Goligher EC, Fan E, Herridge MS, Murray A, Vorona S, Brace D, Rittayamai N, Lanys A, Tomlinson G, Singh JM, Bolz SS, Rubenfeld GD, Kavanagh BP, Brochard LJ, Ferguson ND. Evolution of Diaphragm Thickness during Mechanical Ventilation. Impact of Inspiratory Effort. Am J Respir Crit Care Med. 2015 Nov 1;192(9):1080-8. doi: 10.1164/rccm.201503-0620OC. PMID 26167730
- [Background] Gottesman E, McCool FD. Ultrasound evaluation of the paralyzed diaphragm. Am J Respir Crit Care Med. 1997 May;155(5):1570-4. doi: 10.1164/ajrccm.155.5.9154859.
- [Background] Summerhill EM, El-Sameed YA, Glidden TJ, McCool FD. Monitoring recovery from diaphragm paralysis with ultrasound. Chest. 2008 Mar;133(3):737-43. doi: 10.1378/chest.07-2200. Epub 2008 Jan 15. PMID 18198248
- [Background] Ueki J, De Bruin PF, Pride NB. In vivo assessment of diaphragm contraction by ultrasound in normal subjects. Thorax. 1995 Nov;50(11):1157-61. doi: 10.1136/thx.50.11.1157. PMID 8553271
- [Background] Vivier E, Mekontso Dessap A, Dimassi S, Vargas F, Lyazidi A, Thille AW, Brochard L. Diaphragm ultrasonography to estimate the work of breathing during non-invasive ventilation. Intensive Care Med. 2012 May;38(5):796-803. doi: 10.1007/s00134-012-2547-7. Epub 2012 Apr 5. PMID 22476448
- [Background] Wait JL, Nahormek PA, Yost WT, Rochester DP. Diaphragmatic thickness-lung volume relationship in vivo. J Appl Physiol (1985). 1989 Oct;67(4):1560-8. doi: 10.1152/jappl.1989.67.4.1560. PMID 2676955
- [Background] Matamis D, Soilemezi E, Tsagourias M, Akoumianaki E, Dimassi S, Boroli F, Richard JC, Brochard L. Sonographic evaluation of the diaphragm in critically ill patients. Technique and clinical applications. Intensive Care Med. 2013 May;39(5):801-10. doi: 10.1007/s00134-013-2823-1. Epub 2013 Jan 24. PMID 23344830
- [Background] Noh DK, Lee JJ, You JH. Diaphragm breathing movement measurement using ultrasound and radiographic imaging: a concurrent validity. Biomed Mater Eng. 2014;24(1):947-52. doi: 10.3233/BME-130889. PMID 24211983
- [Background] Scott S, Fuld JP, Carter R, McEntegart M, MacFarlane NG. Diaphragm ultrasonography as an alternative to whole-body plethysmography in pulmonary function testing. J Ultrasound Med. 2006 Feb;25(2):225-32. doi: 10.7863/jum.2006.25.2.225. PMID 16439786
- [Background] Gerscovich EO, Cronan M, McGahan JP, Jain K, Jones CD, McDonald C. Ultrasonographic evaluation of diaphragmatic motion. J Ultrasound Med. 2001 Jun;20(6):597-604. doi: 10.7863/jum.2001.20.6.597. PMID 11400933
- [Derived] Da Conceicao D, Perlas A, Giron Arango L, Wild K, Li Q, Huszti E, Chowdhury J, Chan V. Validation of a novel point-of-care ultrasound method to assess diaphragmatic excursion. Reg Anesth Pain Med. 2024 Nov 4;49(11):800-804. doi: 10.1136/rapm-2023-104983. PMID 37940349